CLINICAL TRIAL: NCT06843187
Title: Lemborexant for the Treatment of Residual Insomnia in Adequately Treated Major Depressive Disorder: a Pilot Randomized Controlled Trial
Brief Title: Lemborexant for the Treatment of Residual Insomnia in Major Depressive Disorder (MDD)
Acronym: MDD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: University of Toronto (Other); Centre for Addiction and Mental Health (Other); Toronto Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 24-133; 68425v4 (Other Grant/Funding Number: Eisai Inc.)
Record Dates: First submitted 2025-01-21; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-09

CONDITIONS: Major Depressive Disorder(MDD); Insomnia Comorbid to Psychiatric Disorder
Keywords: Lemborexant; Residual Insomnia; Major depressive disorder (MDD); Ecological momentary assessments (EMA); Wearable devices; Remote measurement-based care; Randomized controlled trial; Digital health monitoring; Feasibility trial; Pilot study; Placebo-controlled
MeSH Terms: conditions — Depressive Disorder, Major | interventions — lemborexant

STUDY DESIGN:
Intervention Model Description: A double-blind, randomized placebo-controlled pilot trial will be conducted with 30 adults with MDD and residual insomnia. Participants will be randomized to one of two intervention arms (2:1 allocation): lemborexant (experimental group; n = 20) or placebo (control group; n = 10). There will be a 3-week baseline period prior to the 6-week intervention period (lemborexant or a placebo pill for 2 weeks at 5 mg then 4 weeks at 10 mg) and 4-week follow-up period with weekly clinical assessments. Participants will complete a daily digital sleep diary and frequent EMAs on a web-based survey platform as well as passive digital health monitoring via a wearable device. Semi-structured exit interviews will be completed at the end of the study.
Who Masked: Participant, Outcomes Assessor
Masking Description: Data analyst and co-investigators
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lemborexant (Experimental): Participants will take a 5 mg pill of lemborexant daily for two weeks, followed by a dosage increase to 10 mg daily for the next four weeks (6 weeks total).
  Interventions: Drug: Lemborexant
- Placebo (Placebo Comparator): Participants will take a 5 mg of placebo pill daily for 2 weeks then 10 mg daily for 4 weeks (total of 6 weeks).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lemborexant — Dayvigo (lemborexant compound) is an orexin antagonist that acts on the arousal and sleep neural networks of the brain to regulate sleep-wake cycles and is used in the treatment of insomnia characterized by difficulties with sleep.
  Other Names: Dayvigo
  Arms: Lemborexant
Other: Placebo — The placebo is an inactive sugar pill that looks and tastes identical to the lemborexant pill.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if Lemborexant works to treat residual insomnia in adults with depression that is being treated. It will also learn about how practical, tolerable, and effective Lemborexant is. The main questions it aims to answer are:

* Does Lemborexant help participants improve sleep and reduce insomnia symptoms?
* How practical is it to use Lemborexant (how many participants join, drop out, and follow the study rules)? How do participants feel about using it (based on surveys and interviews)?

Researchers will compare Lemborexant to a placebo (a look-alike substance that contains no drug) to see if Lemborexant works to treat residual insomnia in adequately treated major depressive disorder.

Participants will:

* Take Lemborexant or a placebo every day for 6 weeks (2 weeks at 5 mg then 4 weeks at 10 mg)
* Complete clinical assessments and in-person study visits
* Maintain a digital sleep diary and complete daily and weekly self-report ecological momentary assessments (EMAs)
* Use a wearable device which will be used to collect and monitor physiological data

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is often accompanied by persistent residual insomnia which does not resolve, even after adequate MDD treatment. Lemborexant is an orexin receptor antagonist involved in the regulation of sleep-wake cycles with a favourable safety profile compared to other sleep medications. There are currently no trials evaluating the feasibility and clinical efficacy of Lemborexant as a treatment for residual insomnia in patients with adequately treated MDD. This pilot study will investigate the feasibility, tolerability, and efficacy of Lemborexant in adults with adequately-treated MDD and residual insomnia.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 70 (inclusive), with a self-reported body mass index (BMI) between 19 and 35 kg/m2 (inclusive).
2. Meet criteria for MDD without psychotic symptoms as defined by the Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM-5) and currently in a MDE as confirmed by the MINI International Neuropsychiatric Interview (MINI).
3. Have not failed more than 2 trials of antidepressant treatments in the current MDE, and have a history of adequate response (clinical outcome rating score of 1 or 2) to at least 1 antidepressant treatment during the current MDE as determined by the Antidepressant Treatment History Form-Short Form (ATHF-SF).
4. Are outpatients.
5. Did not take non-psychotropic or non-central nervous system (CNS) medications suspected to affect sleep-wake function for at least 4 weeks before starting the study.
6. At screening visit 1, self-reported subjective total sleep time (sTST) ≤ 6.5 hours, subjective sleep onset latency (sSOL) ≥ 30 mins, and subjective wake time after sleep onset (sWASO) ≥ 45 mins per night at least three times per week 1 month prior to screening.
7. At screening visit 1, self-reported regular time spent in bed, either sleeping or trying to sleep must be between 7 and 10 hours, inclusive.
8. At screening visit 1, self-reported regular bedtime (i.e., the time the participant gets in bed) between 21:00 and 01:00 and regular wake time (i.e., the time participant wakes and does not go back to sleep) between 05:00 and 10:00.
9. At screening visit 2, confirmation of current insomnia symptoms as determined from responses on the Sleep Diary completed on at least 7 consecutive mornings (minimum 5 of 7 for eligibility), such that sSOL ≥ 30 mins on at least 3 of the 7 nights and/or sWASO ≥ 45 mins on at least 3 of the 7 nights.
10. At screening visit 2, confirmation of sufficient duration of time spent in bed, as determined from responses on the Sleep Diary on the 7 most recent mornings before the visit, such that there are no more than 2 nights with time spent in bed of duration < 7 hours or > 10 hours.
11. At screening visit 2, confirmation of regular bedtime (i.e., the time the participant gets in bed) between 21:00 and 01:00 on at least 5 of the 7 preceding nights, and regular wake time (i.e., the time the participant wakes and does not go back to sleep) between 05:00 and 10:00 on at least 5 of the 7 preceding nights.
12. Are able to understand and comply with the requirements of the study, as judged by the investigator(s).
13. Provide written informed consent before initiation of any study-related procedures.
14. Own a smartphone and have reliable access to the internet and a browser on which to complete questionnaires.

Exclusion Criteria:

1. Previously participated in any clinical trial of lemborexant.
2. Have any known sensitivity to lemborexant or their excipients.
3. Failed treatment with an appropriate dose or adequate duration of dual orexin receptor antagonist drugs (efficacy or safety), in the opinion of the investigator.
4. Women who are pregnant or lactating (documented by a positive beta-human chorionic gonadotropin [beta-hCG] or human chorionic gonadotropin [hCG] urine test with a minimum sensitivity of 25 IU/L or equivalent units of beta-hCG or hCG).
5. Women who are not using any of the following approved and effective method of contraception or family planning during the study: Combined estrogen- and progestogen-containing hormonal contraception associated with inhibition of ovulation (oral, intravaginal, or transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, or implantable), intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion and litigation, vasectomized partner, sexual abstinence, or two forms of contraception with any barrier method or oral hormones (e.g., condom plus diaphragm, condom or diaphragm plus spermicide, oral hormonal contraceptives plus spermicide or condom).
6. If participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions or the therapeutic focus 4 weeks before screening and the entire duration of participation.
7. Unable to keep any current psychiatric medications unchanged for 4 weeks before screening and for the entire duration of participation in the study.
8. Have active suicidal intent as determined by a score of 3 (severe suicidality with a clear plan and/or intent) or 4 (very severe: suicidal attempts) on item #3 on the HAM-D-17.
9. Have had a course of electroconvulsive therapy or intravenous ketamine therapy in the current episode or any previous episode.
10. According to medical history, have had insomnia associated with another sleep disorder or have a history of any condition that impacted or was likely to impact sleep, including any lifetime diagnosis of sleep-related breathing disorder, periodic limb movement disorder, restless legs syndrome, nightmare disorder, sleep terror disorder, sleepwalking disorder, rapid eye movement (REM) behaviour disorder, or narcolepsy.
11. Exclusionary score on screening instruments to rule out individuals with symptoms of certain sleep disorders other than insomnia: Snoring, Tiredness, Observed Apnea, High Blood Pressure, BMI, Age, Neck circumference, and Gender (STOP-Bang) scores ≥ 5; International Restless Legs Scale (IRLS) scores ≥ 16, Epworth Sleepiness Scale (ESS) > 15.
12. Habitual naps during the day more than 3 times/week.
13. Transmeridian travel across more than 3 time zones in the 2 weeks before screening, or between screening and study baseline, or plans to travel across more than 3 time zones during the study.
14. Used any modality of treatment for insomnia, including cognitive-behavioural therapy or cannabis within 2 weeks before screening.
15. Excessive caffeine use that in the opinion of the investigator contributes to the participant's insomnia, or habitually consumes caffeine-containing beverages after 18:00.
16. Reports habitually consuming more than 14 drinks containing alcohol per week (females) or more than 21 drinks containing alcohol per week (males).
17. Used prohibited prescriptions or over-the-counter concomitant medications, or used any medication or sleep aid with known effects on sleep within 2 weeks before screening.
18. Comorbid nocturia that is causing or exacerbating the insomnia.
19. Report a history of sleep-related violent behaviour, or sleep driving, or any other complex sleep-related behaviour (e.g., making phone calls, preparing and eating food).
20. Report symptoms potentially related to narcolepsy that in the clinical opinion of the investigator indicates the need for a diagnostic referral for the presence of narcolepsy.
21. For participants who underwent polysomnography (PSG) within the previous year before informed consent:

    1. Age 18-64 years old, inclusive: Apnea Hypopnea Index ≥ 10, or Periodic Limb Movement with Arousal Index ≥ 10.
    2. Age ≥ 65 years old: Apnea Hypopnea Index > 15, or Periodic Limb Movement with Arousal Index > 15.
22. Diagnosis of substance dependence or abuse within the last 3 months as determined by MINI.
23. Lifetime history of bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or current psychotic symptoms as determined by MINI.
24. Have a MINI diagnosis of obsessive-compulsive disorder, post-traumatic stress disorder (current), assessed by a study investigator to be primary and causing greater impairment than MDD.
25. Have a diagnosis of any personality disorder that is assessed by a study investigator to be primary and causing greater impairment than MDD.
26. Have a concomitant major unstable medical illness, cardiac pacemaker, or implanted medication pump.
27. Have any significant neurological disorder or insult including, but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, any history of seizure except a febrile seizure of infancy, cerebral aneurysm, Parkinson's disease, Huntington's chorea, multiple sclerosis, significant head trauma with loss of consciousness for greater than 5 minutes.
28. A history of risk factors for Torsade de Pointes (e.g., heart failure, hypokalemia, family history of long QT syndrome) or the use of concomitant medications that prolonged the QTcF interval.
29. Scheduled for major surgery during the study.
30. Have a clinical finding that is unstable or that, in the opinion of the investigator(s), would be negatively affected by the study medication or that would affect the study medication (e.g., diabetes mellitus, hypertension, unstable angina).
31. Have uncorrected hypothyroidism or hyperthyroidism. Subjects needing a thyroid hormone supplement to treat hypothyroidism must have been on a stable dose of the medication for 30 days prior to enrolment.
32. Have any other condition that, in the opinion of the investigator(s), would adversely affect the subject's ability to complete the study or its measures.
33. Justifications for any exclusions based on race, gender, or ethnicity: Non-English-speaking individuals are excluded because the ability to communicate study information, answer questions accurately and completely about the study, and obtain consent are necessary.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility Outcomes | 13 weeks
  Feasibility will be measured by the recruitment rate, withdrawal rate, data completion rate, and adherence rate. Recruitment rate will be quantified by the percentage of eligible participants enrolled relative to the number of participants contacted. Feasibility will be marked as a minimum of 1-2 participants enrolled per month. Withdrawal/dropout rate will be quantified by the percentage of participants who drop out of the study. The upper limit of the 95% confidence interval (CI) for dropout rate should not exceed 20%.
  Adherence and data completion will bhe proportion of participants who strictly follow the study protocol (the "per-protocol group") will be estimated with a 95% CI. This includes adherence to treatment (taking the medication correctly for six weeks), study completion (attending all required visits), and providing complete data. To be considered feasible, the lower limit of this 95% CI must be greater than 80%.
Tolerability Outcomes | 10 weeks
  Tolerability will be measured by the frequency and nature of adverse events and medication adherence (i.e., missed dosage).

SECONDARY OUTCOMES:
Preliminary Clinical Parameters | 6 weeks
  Changes in insomnia symptoms will be measured using the Insomnia Severity Index (ISI) Score. ISI score reduction will be compared between allocation and treatment end for participants randomized to receive Lemborexant and those receiving placebo.
Within-person Correlations | 10 weeks
  Within-person changes in insomnia symptoms will be measured by within-person correlations of baseline and follow-up ISI scores. The ISI assesses the severity of insomnia symptoms, such as the impact of sleep on daytime functioning, difficulties with sleep onset, and sleep maintenance. Each item is rated on a scale from 0 (mild) to 4 (very severe), with a higher overall score indicating more severe insomnia presentations.
Standard Deviation | 13 weeks
  Within and between participant variability in insomnia symptoms will be measured by standard deviation of ISI scores. This measure will be separate for each group (treatment and placebo).
Change in Physiological Biometrics (Oura Ring Metrics) | 13 weeks
  Physiological biometrics will be captured using the Oura Ring and analyzed as a composite measure of changes across multiple parameters. Individual metrics will be reported separately and summarized as part of an overall physiological profile. The measured parameters include daily activity (step count (steps/day) and energy expenditure (METs)), heart rate metrics (resting heart rate (beats per minute) and heart rate variability (milliseconds)), body temperature (average nightly body temperature deviation (degrees Celsius), sleep quality (sleep latency, total time in bed, sleep staging (light, deep, REM sleep in minutes)), wake onset (minutes), and Oura composite scores (sleep, activity, and readiness scores (0-100 scale)). Statistical analyses will assess changes in each metric individually, as well as aggregated trends across sleep, activity, and recovery domains.
Patient Health Questionnaire-9 (PHQ-9) | 13 weeks
  This questionnaire assesses the severity of depression, with questions probing the frequency and severity of symptoms such as mood, energy, sleep, and concentration. Each item is scored from 0 (not at all) to 3 (nearly every day), with a higher total score indicating more severe depression presentations.
Insomnia Severity Index (ISI-7) | 13 weeks
  This questionnaire assesses the severity of insomnia symptoms, such as the impact of sleep on daytime functioning, difficulties with sleep onset, and sleep maintenance. Each item is rated on a scale from 0 (mild) to 4 (very severe), with a higher overall score indicating more severe insomnia presentations.
Generalized Anxiety Disorder-7 (GAD-7) | 13 weeks
  This questionnaire assesses the severity of anxiety symptoms, such as excessive worry, restlessness, and irritability. Each question is scored ranging from 0 (not at all) to 3 (nearly every day), with a higher overall score indicating more severe presentations of anxiety.
World Health Organization Well-being Index (WHO-5) | 13 weeks
  This questionnaire is a self-report measure that evaluates subjective well-being, with statements probing mood, vitality, and mental well-being. Participants rate their responses from 0 (at no time) to 5 (all the time), with a higher overall score indicating positive well-being.
Montgomery-Åsberg Depression Rating Scale (MADRS) | 13 weeks
  This clinician-administered scale assesses the severity and changes in depression symptoms over time. Each item is rated from 0 (no symptoms) to 6 (very severe symptoms), with a higher overall score indicating more severe depression.

OTHER OUTCOMES:
Patient Perspectives | 13 weeks
  Subjective patient experiences, thoughts, beliefs, and attitudes towards the digital health monitoring platforms (REDCap and Oura Ring) will be assessed using the user experience survey and semi-structured exit interviews. Open-ended feedback for considerations of future trials and digital intervention design will be considered.

CONTACTS AND LOCATIONS:
Overall Officials: Venkat Bhat, MD, MSc, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Unity Health Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manual (on) Transcription: Transcription Conventions, Software Guides and Practical Hints for Qualitative Researchers. 3. Engl. Ed., January 2015. Marburg: dr. dresing et pehl GmbH; 2015.
- [Background] Wilson EB. Probable Inference, the Law of Succession, and Statistical Inference. J Am Stat Assoc. 1927;22: 209-212. doi:10.1080/01621459.1927.10502953
- [Background] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Bang H, Flaherty SP, Kolahi J, Park J. Blinding assessment in clinical trials: A review of statistical methods and a proposal of blinding assessment protocol. Clin Res Regul Aff. 2010;27: 42-51. doi:10.3109/10601331003777444
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Edward KL, Garvey L, Aziz Rahman M. Wearable activity trackers and health awareness: Nursing implications. Int J Nurs Sci. 2020 Mar 25;7(2):179-183. doi: 10.1016/j.ijnss.2020.03.006. eCollection 2020 Apr 10. PMID 32685614
- [Background] Lee S, Kim H, Park MJ, Jeon HJ. Current Advances in Wearable Devices and Their Sensors in Patients With Depression. Front Psychiatry. 2021 Jun 17;12:672347. doi: 10.3389/fpsyt.2021.672347. eCollection 2021. PMID 34220580
- [Background] Ahmed A, Aziz S, Alzubaidi M, Schneider J, Irshaidat S, Abu Serhan H, Abd-Alrazaq AA, Solaiman B, Househ M. Wearable devices for anxiety & depression: A scoping review. Comput Methods Programs Biomed Update. 2023;3:100095. doi: 10.1016/j.cmpbup.2023.100095. Epub 2023 Jan 30. PMID 36743720
- [Background] Martin J, Rueda A, Lee GH, Tassone VK, Park H, Ivanov M, Darnell BC, Beavers L, Campbell DM, Nguyen B, Torres A, Jung H, Lou W, Nazarov A, Ashbaugh A, Kapralos B, Litz B, Jetly R, Dubrowski A, Strudwick G, Krishnan S, Bhat V. Digital Interventions to Understand and Mitigate Stress Response: Protocol for Process and Content Evaluation of a Cohort Study. JMIR Res Protoc. 2024 May 6;13:e54180. doi: 10.2196/54180. PMID 38709554
- [Background] Eisai Inc. PRODUCT MONOGRAPH INCLUDING PATIENT MEDICATION INFORMATION: DAYVIGO Lemborexant Tablet Tablet, 5 mg, 10 mg, Oral. 2023.
- [Background] Uzun S, Kozumplik O, Jakovljevic M, Sedic B. Side effects of treatment with benzodiazepines. Psychiatr Danub. 2010 Mar;22(1):90-3. PMID 20305598
- [Background] Yardley J, Karppa M, Inoue Y, Pinner K, Perdomo C, Ishikawa K, Filippov G, Kubota N, Moline M. Long-term effectiveness and safety of lemborexant in adults with insomnia disorder: results from a phase 3 randomized clinical trial. Sleep Med. 2021 Apr;80:333-342. doi: 10.1016/j.sleep.2021.01.048. Epub 2021 Feb 1. PMID 33636648
- [Background] Eisai Inc. U.S. FDA APPROVES EISAI'S DAYVIGOTM (LEMBOREXANT) FOR TREATMENT OF INSOMNIA IN ADULT PATIENTS. 2019. Available: https://www.eisai.com/news/2019/news201993.html#:~:text=IN%20ADULT%20PATIENTS-,U.S.%20FDA%20APPROVES%20EISAI'S%20DAYVIGO%E2%84%A2%20(LEMBOREXANT)%20FOR%20TREATMENT%20OF,OF%20MORE%20THAN%202%2C000%20PATIENTS
- [Background] Regulatory Decision Summary for Dayvigo. Government of Canada; 2024. Available: https://dhpp.hpfb-dgpsa.ca/review-documents/resource/RDS00757
- [Background] Nakamura M, Nagamine T. Neuroendocrine, Autonomic, and Metabolic Responses to an Orexin Antagonist, Suvorexant, in Psychiatric Patients with Insomnia. Innov Clin Neurosci. 2017 Apr 1;14(3-4):30-37. eCollection 2017 Mar-Apr. PMID 28584695
- [Background] Kuriyama A, Tabata H. Suvorexant for the treatment of primary insomnia: A systematic review and meta-analysis. Sleep Med Rev. 2017 Oct;35:1-7. doi: 10.1016/j.smrv.2016.09.004. Epub 2016 Oct 28. PMID 28365447
- [Background] Michelson D, Snyder E, Paradis E, Chengan-Liu M, Snavely DB, Hutzelmann J, Walsh JK, Krystal AD, Benca RM, Cohn M, Lines C, Roth T, Herring WJ. Safety and efficacy of suvorexant during 1-year treatment of insomnia with subsequent abrupt treatment discontinuation: a phase 3 randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2014 May;13(5):461-71. doi: 10.1016/S1474-4422(14)70053-5. Epub 2014 Mar 27. PMID 24680372
- [Background] Triantafillou S, Saeb S, Lattie EG, Mohr DC, Kording KP. Relationship Between Sleep Quality and Mood: Ecological Momentary Assessment Study. JMIR Ment Health. 2019 Mar 27;6(3):e12613. doi: 10.2196/12613. PMID 30916663
- [Background] Fortuyn HA, Lappenschaar MA, Furer JW, Hodiamont PP, Rijnders CA, Renier WO, Buitelaar JK, Overeem S. Anxiety and mood disorders in narcolepsy: a case-control study. Gen Hosp Psychiatry. 2010 Jan-Feb;32(1):49-56. doi: 10.1016/j.genhosppsych.2009.08.007. Epub 2009 Oct 1. PMID 20114128
- [Background] Grafe LA, Bhatnagar S. Orexins and stress. Front Neuroendocrinol. 2018 Oct;51:132-145. doi: 10.1016/j.yfrne.2018.06.003. Epub 2018 Jun 19. PMID 29932958
- [Background] Salomon RM, Ripley B, Kennedy JS, Johnson B, Schmidt D, Zeitzer JM, Nishino S, Mignot E. Diurnal variation of cerebrospinal fluid hypocretin-1 (Orexin-A) levels in control and depressed subjects. Biol Psychiatry. 2003 Jul 15;54(2):96-104. doi: 10.1016/s0006-3223(02)01740-7. PMID 12873798
- [Background] Schmidt FM, Brugel M, Kratzsch J, Strauss M, Sander C, Baum P, Thiery J, Hegerl U, Schonknecht P. Cerebrospinal fluid hypocretin-1 (orexin A) levels in mania compared to unipolar depression and healthy controls. Neurosci Lett. 2010 Oct 8;483(1):20-2. doi: 10.1016/j.neulet.2010.07.038. Epub 2010 Jul 22. PMID 20655364
- [Background] Brundin L, Bjorkqvist M, Petersen A, Traskman-Bendz L. Reduced orexin levels in the cerebrospinal fluid of suicidal patients with major depressive disorder. Eur Neuropsychopharmacol. 2007 Sep;17(9):573-9. doi: 10.1016/j.euroneuro.2007.01.005. Epub 2007 Mar 7. PMID 17346943
- [Background] Nollet M, Leman S. Role of orexin in the pathophysiology of depression: potential for pharmacological intervention. CNS Drugs. 2013 Jun;27(6):411-22. doi: 10.1007/s40263-013-0064-z. PMID 23657787
- [Background] Nollet M, Gaillard P, Tanti A, Girault V, Belzung C, Leman S. Neurogenesis-independent antidepressant-like effects on behavior and stress axis response of a dual orexin receptor antagonist in a rodent model of depression. Neuropsychopharmacology. 2012 Sep;37(10):2210-21. doi: 10.1038/npp.2012.70. Epub 2012 Jun 20. PMID 22713907
- [Background] Nollet M, Gaillard P, Minier F, Tanti A, Belzung C, Leman S. Activation of orexin neurons in dorsomedial/perifornical hypothalamus and antidepressant reversal in a rodent model of depression. Neuropharmacology. 2011 Jul-Aug;61(1-2):336-46. doi: 10.1016/j.neuropharm.2011.04.022. Epub 2011 Apr 23. PMID 21530551
- [Background] Scammell TE. Narcolepsy. N Engl J Med. 2015 Dec 31;373(27):2654-62. doi: 10.1056/NEJMra1500587. No abstract available. PMID 26716917
- [Background] Yoshida Y, Fujiki N, Nakajima T, Ripley B, Matsumura H, Yoneda H, Mignot E, Nishino S. Fluctuation of extracellular hypocretin-1 (orexin A) levels in the rat in relation to the light-dark cycle and sleep-wake activities. Eur J Neurosci. 2001 Oct;14(7):1075-81. doi: 10.1046/j.0953-816x.2001.01725.x. PMID 11683899
- [Background] Pae CU, Tharwani H, Marks DM, Masand PS, Patkar AA. Atypical depression: a comprehensive review. CNS Drugs. 2009 Dec;23(12):1023-37. doi: 10.2165/11310990-000000000-00000. PMID 19958040
- [Background] Alijanpour S, Khakpai F, Ebrahimi-Ghiri M, Zarrindast MR. Co-administration of the low dose of orexin and nitrergic antagonists induces an antidepressant-like effect in mice. Biomed Pharmacother. 2019 Jan;109:589-594. doi: 10.1016/j.biopha.2018.10.033. Epub 2018 Nov 3. PMID 30399595
- [Background] Berridge CW, Espana RA. Hypocretins: waking, arousal, or action? Neuron. 2005 Jun 2;46(5):696-8. doi: 10.1016/j.neuron.2005.05.016. PMID 15924855
- [Background] Nutt D, Wilson S, Paterson L. Sleep disorders as core symptoms of depression. Dialogues Clin Neurosci. 2008;10(3):329-36. doi: 10.31887/DCNS.2008.10.3/dnutt. PMID 18979946
- [Background] Shariq AS, Rosenblat JD, Alageel A, Mansur RB, Rong C, Ho RC, Ragguett RM, Pan Z, Brietzke E, McIntyre RS. Evaluating the role of orexins in the pathophysiology and treatment of depression: A comprehensive review. Prog Neuropsychopharmacol Biol Psychiatry. 2019 Jun 8;92:1-7. doi: 10.1016/j.pnpbp.2018.12.008. Epub 2018 Dec 18. PMID 30576764
- [Background] Health Quality Ontario. Psychotherapy for Major Depressive Disorder and Generalized Anxiety Disorder: A Health Technology Assessment. Ont Health Technol Assess Ser. 2017 Nov 13;17(15):1-167. eCollection 2017. PMID 29213344